CLINICAL TRIAL: NCT06265298
Title: Implementation of a Protocol for the Transdifferentiation of Buccal Mucosal Epithelium Into Corneal Epithelium
Acronym: TransBuCor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institute for Neuroscience Montpellier (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL23_0099
Record Dates: First submitted 2024-01-24; First posted 2024-02-20 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Limbal Stem Cell Deficiency
Keywords: epithelium; mucosa; cornea; corneal epithelium
MeSH Terms: conditions — Limbal Stem Cell Deficiency; Corneal Diseases

STUDY DESIGN:
Intervention Model Description: transversal and fundamental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reconstruction conjonctival (Experimental): Patients undergoing conjunctival reconstruction using oral mucosa
  Interventions: Procedure: Conjunctival reconstruction

INTERVENTIONS:
Procedure: Conjunctival reconstruction — Conjunctival reconstruction using buccal mucosa taken from the patient's mouth. Following the reconstruction operation, an additional biopsy of buccal mucosa will be taken to develop a laboratory protocol for the transdifferentiation of these buccal cells into corneal epithelial stem cells.

SUMMARY:
Objectives The transparent surface of the eye, called the cornea, plays a crucial role in transmitting light to the retina and in protecting the eye. On its external surface, the cornea is composed of a constantly renewing multistratified epithelium. This mechanism is fueled by stem cells located in the limbus (the transition zone between the cornea and the sclera). Limbal Stem Cell Deficiency (LSCD) is characterized by a decrease or cessation of epithelial renewal and neovascularization of the cornea. Consequently, the cornea loses its integrity and transparency. This visually impairing condition is currently in a therapeutic impasse as only autologous limbal or allogeneic corneal grafts are viable options, but they pose significant risks to patients.

Studies have shown that the oral cavity contains stem cells that can be isolated, cultured, and transdifferentiated into limbal stem cells (LSCs). However, to date, these studies are limited, and no protocol has been validated. In this study, the advantage of the accessibility of the oral cavity is used to develop a protocol for differentiating cells from the oral mucosa into limbal stem cells (LSCs) for use in a future clinical trial with patients.

Methodology This prospective monocentric study will be conducted on patients from the ophthalmology department of the Montpellier University Hospital who have an indication for conjunctival reconstruction. After obtaining consent from the patients, cells from the oral wall will be sent to the tissue bank of the Montpellier University Hospital, where they will be cultured. Finally, the transdifferentiation steps will be analyzed by the "Eye" research team at the Institute of Neuroscience in Montpellier, which is collaborating on the project. The investigators have established objective factors to assess the success of the developed protocol based on the literature : (i) > 3% of stem cells in primary cultures, (ii) <10% aborted colonies, (iii) Expression of LSC markers (Pax6, Krt14, p63).

DETAILED DESCRIPTION:
1. Recall on Corneal Anatomy and Histology

   The cornea is an essential ocular component for vision: often referred to as the first "transparent porthole" at the front of the eye. It is the first structure that light encounters upon entering the eye. Its primary role is to converge incident light rays, which then proceed towards the lens before reaching the retina and initiating the visual cascade.

   The cornea is an avascular and transparent tissue composed of five layers: corneal epithelium, Bowman's layer, corneal stroma, Descemet's membrane, and corneal endothelium.
   * The corneal epithelium is the outermost layer of the cornea, consisting of corneal epithelial cells, accounting for about 10% of the entire cornea. This layer constantly regenerates, with complete renewal occurring every seven days. Scratches on this layer generally heal well.
   * The Bowman's layer helps bind the corneal epithelium and stroma together. This layer cannot regenerate once damaged, potentially leading to permanent scars that can affect vision.
   * The corneal stroma represents about 90% of the cornea and is composed of collagen and keratocytes.
   * Descemet's membrane is made up of collagen and separates the corneal stroma from the endothelium. This layer gradually thickens with age.
   * The corneal endothelium is the innermost layer and aids in transporting fluid from other corneal layers. Damage to this layer can compromise this process and negatively impact a person's vision.
2. Renewal and Healing Process of Corneal Epithelium

   Corneal epithelial cells regenerate within 3 to 10 days through constant renewal from limbal stem cells located at the limbus (transition zone between the cornea and sclera) in the basal cell layer, within pigmented crypts called Vogt's palisades.

   Deficiency In Limbal Stem Cells (LSCD) is characterized by a loss or impairment of limbal stem cells crucial for corneal epithelial repopulation and limbal barrier function.

   The etiologies of LSCD can be genetic (PAX6), secondary to chronic inflammation (e.g., severe allergic keratoconjunctivitis or ocular rosacea), acquired through infection such as herpetic keratitis, or secondary to a blistering disease such as Steven-Johnson syndrome or Lyell syndrome. LSCD can also be acquired through trauma from chemical or thermal burns. Etiologies can also be idiopathic.

   When these stem cells are lost, the corneal epithelium is unable to repair and renew itself. This leads to epithelial degradation, persistent epithelial defects, conjunctivalization, corneal neovascularization, corneal scars, and chronic inflammation. These factors contribute to photophobia, loss of corneal clarity, vision loss, and chronic pain. This makes corneal transplantation impossible as it would be rejected and/or exhibit poor healing.

   Current solutions for addressing this cause of corneal blindness are limited. Techniques include autologous limbal grafts from the patient's contralateral eye, but this may pose risk and is not possible when the pathology is bilateral. Allogeneic grafts are highly risky for rejection and require systemic immunosuppressive treatment.
3. Mucous Membrane Grafts in Periorbital Reconstruction

Oral mucosa grafting is a well-established surgical technique for treating conjunctival deficiencies and scars. Oral mucosa possesses biological properties similar to conjunctiva, both being composed of one or more layers of epithelial cells covering a loose connective tissue layer. It can be harvested repeatedly, with the donor site easily accessible and widely available. Donor site morbidity is low, and surgery is generally well-tolerated by patients. Moreover, the surgical technique is relatively simple, making oral mucosa an ideal candidate for replacing conjunctival anomalies.

Oral mucosa grafts have been used not only for treating contracted sockets in anophthalmic patients and reconstructing the ocular surface and fornix in patients after tumor resection but also for treating refractive pterygium and in patients with pemphigoid or ocular symblepharon. It is also the most commonly used tissue in treating post-surgical complications, including conjunctival deficiencies after glaucoma, retinal surgery, corneal melts related to keratoprosthesis, and covering the dacryocystorhinostomy tract. Additionally, oral mucosa has been used to repair intractable sclerocorneal melts caused by severe chemical burns.

Some teams have proposed using buccal mucosa cells and transdifferentiating them into limbal stem cells. The oral cavity is easily accessible, and stem cells can be isolated from the mucosa in a minimally invasive and low-risk manner for the patient. These cells have a high differentiation potential and express markers of embryonic stem cells; Tra2-49, Tra2-54, SSEA4, Oct4, Sox2, and Nanog, as well as the neural crest marker Nestin. However, human trials are still in the preliminary stage, and no therapy has been validated to date.

In this proof-of-concept study, the aim is to develop a protocol for differentiating oral mucosa cells into limbal stem cells for use in a future clinical trial with patients.

ELIGIBILITY:
Inclusion Criteria:

* Presenting an indication for conjunctival reconstruction using oral mucosa (for example because of a recurrent pterygium, conjunctival carcinoma or ocular burn)
* Written consent to participate in this research

Exclusion Criteria:

* Chronic infection (HIV, hepatitis, tuberculosis, Lyme disease)
* Oral pathology which could affect the health of the oral mucosa tissue according to the opinion of the investigating doctor
* Uncontrolled systemic disease
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Successful Transdifferentiation | change over time between Baseline and 14 days
  Successful differentiation, defined by the percentage of stem cells on primary cultures ≥ 3%
Successful Transdifferentiation | change over time between Baseline and 14 days
  Successful differentiation, defined by the percentage of aborted colonies < 10%.
Successful Transdifferentiation | change over time between Baseline and 14 days
  The quantitative real-time polymerase chain reaction, (qPCR) technique will be used to monitor expression levels of limbal stem cell markers such as Krt14 and Krt5.
  The qPCR technique will be used to monitor expression levels of transcription factors.
Successful Transdifferentiation | change over time between Baseline and 14 days
  Successful differentiation, defined by the presence of transcription factors p63 and Pax6
  The qPCR technique will be used to monitor expression levels of transcription factors.
Successful Transdifferentiation | change over time between Baseline and 14 days
  The qPCR technique will be used wiil be used to monitor the absence of expression of markers of terminal differentiation of corneal epithelial cells, such as Krt3 and Krt12

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Daien, MD PhD, Study Director — v-daien@chu-montpellier.fr
Locations (1):
- CHU Gui de Chauliac - Service d'Ophtamologie, Montpellier, Occitanie, France

IPD SHARING:
Plan to Share IPD: No